CLINICAL TRIAL: NCT05494931
Title: Effect of Superficial Keratotomy on Reducing Postoperative Pain Fallowing Conjuctival Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasser Karimi, Principal Investigator, Assistant Professor, Iran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR.IUMS.FMD.REC.1401.021
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Reduced Corneal Sensation
Keywords: keratotomy.conjuctival flap.radial corneal nerve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In this first group, the same classic method of Gunderson conjunctival flap surgery will be used.
- intervention group (Active Comparator): in the this group, Gunderson conjunctival flap surgery will be performed adjuncted by corneal neurotomy
  Interventions: Procedure: corneal neurotomy

INTERVENTIONS:
Procedure: corneal neurotomy — Classic Gunderson conjunctival flap surgery adjuncted by corneal neurotomy
  Arms: intervention group

SUMMARY:
During conjunctival flap surgery the corneal epithelium is removed and a conjunctival flap is placed on the cornea and after a few weeks the conjunctiva covers the surface of the eye.

Complications of this operation are flap retraction, conjunctival inclusion cysts, bleeding, infection and pain. Pain is one of the main complications of conjunctival flap surgery. Two sources are conceivable for pain: 1) conjunctival pain 2) corneal pain, the second of which is the main part of the pain.

Numerous methods for controlling corneal pain have been reported in various articles. Eye patches are often recommended for the treatment of corneal abrasions despite the lack of evidence. Recommended analgesics to control corneal scratch pain include nonsteroidal anti-inflammatory drugs (NSAIDs), local anesthetics, and topical cycloplegias.

In this article, we are going to review and evaluate a new method called corneal neuorotomy, i.e., corneal nerve endings that inserted radially can be cut to reduce postoperative pain.

DETAILED DESCRIPTION:
The main idea of this randomized clinical trial is to test the extent of pain relief after incision of radial corneal nerve endings.

Patients are divided into two groups. In the first group, the same classic method of conjunctival flap surgery was used and in the second group, conjunctival flap surgery was performed adjuncted by cutting the radial superficial nerves of the cornea. The postoperative pain scores of these two groups will be measured using visual analogue scale, after 6 hours, 24 hours and 48 hours, and finally the average pain of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* VLE (vision loss eye)Patients who are candidates for prosthesis implantation

Exclusion Criteria:

* 1 painful vision loss eye
* 2 Patients who are candidates for conjunctival flap with indications other than implant placement (such as pain due to corneal ulcers, etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
postoperative pain 6 hours after conjunctival flap | 6 hours after surgery
  measured via self-reported visual analogue scale (0 -10) , higher score means more severe pain
postoperative pain 24 hours after conjunctival flap | 24 hours after surgery
  measured via self-reported visual analogue scale (0 -10) , higher score means more severe pain
postoperative pain 48 hours after conjunctival flap | 48 hours after surgery
  measured via self-reported visual analogue scale (0 -10) , higher score means more severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Center, Tehran, Tehrani, Iran